CLINICAL TRIAL: NCT00614224
Title: Structural Neuroplasticity Associated With Aerobic Treadmill Training in Geriatric Chronic Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andreas R Luft (Other)
Collaborators: Robert Bosch Medical Center (Other); Max-Planck-Institute Tuebingen (Other)
Responsible Party: Sponsor-Investigator, Andreas R Luft, Prof, University Hospital Tuebingen
Organization: University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOSCH-TAEX-001
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2008-01

CONDITIONS: Stroke; Hemiparesis
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Treadmill training group (TAEX)
  Interventions: Behavioral: treadmill exercise training
- B (Active Comparator): Attention control group (CON)
  Interventions: Behavioral: treadmill exercise training

INTERVENTIONS:
Behavioral: treadmill exercise training — 3 months (3 times/week) progressive graded aerobic treadmill training with a duration of 10-45 min per training session

SUMMARY:
Aerobic treadmill exercise has been shown to improve walking, cardiovascular fitness and thereby risk factor profiles in chronic stroke patients (Macko et al., Stroke 2005). The proposed project is a randomized controlled trial in geriatric stroke patients with chronic disabilities to investigate potential mechanisms of treadmill therapy. The hypothesis is tested that 3-months of aerobic treadmill exercise induces structural brain plasticity and reorganization. The outcome measures are walking ability, gait pattern, cardiovascular fitness and brain morphology. This study will elucidate fundamental mechanisms of brain adaptations linked to task-repetitive aerobic lower extremity exercise. These mechanisms will not only lead to a better understanding but may also help to identify predictors of treatment response.

40 patients aged over 60 years with lower extremity paresis after a first-ever clinical stroke longer than 6 months prior to study inclusion will be recruited from: 1) The Geriatric Rehabilitation Clinic at the Robert-Bosch Hospital in Stuttgart 2) the Dept of Neurology, University Hospital in Tübingen. Subjects will be randomized to 3 months progressive graded aerobic treadmill exercise training (TAEX; 3 times/week, duration 10-45 min) or an attention control group (CON). Because we expect that localization and size of stroke affect therapy outcomes, stratified randomization will be used to balance entry into groups.

We hypothesize that 3 months of treadmill gait training but not conventional care leads to improvements of cardiovascular fitness and gait and to brain reorganization (structural plasticity) in regions in which functional adaptations have been demonstrated using fMRI in previous studies. The specific aims are:

* To assess reorganization by comparing cortical thickness, cortical density and fiber tract morphology before (time point 0), and after therapy (3 months) using T1-weighted 3D-MPRAGE images, voxel based morphometry and diffusion tensor imaging.
* To correlate brain reorganization with improvements in walking velocity, and analysis of gait patterns (parameters, swing time, stance time, gait symmetry).
* To correlate brain reorganization with location and size of the index stroke lesion and of diffuse white matter damage (subcortical vascular encephalopathy). Lesion and white matter damage will be evaluated based on T2-weighted FLAIR sequences.

ELIGIBILITY:
Inclusion Criteria:

* women and men aged > 60 years
* first ever ischemic stroke at least prior 6 months
* all conventional inpatient and outpatient physical therapy completed
* residual hemiparetic gait disturbance adequate language and neurocognitive function to participate in exercise training and testing

Exclusion Criteria:

* already performing > 20 minutes aerobic exercise 3 X/ week
* Alcohol consumption >2 oz liquor, or 2x 4oz glasses of wine, or 2x 12 oz cans of beer per day.
* Cardiac history of

  1. unstable angina
  2. recent (< 3 months) myocardial infarction
  3. congestive heart failure (NYHA category II)
  4. hemodynamically significant valvular dysfunction.
* Medical History:

  1. recent hospitalization (<3 months) for severe medical disease
  2. symptomatic peripheral arterial occlusive disease
  3. orthopedic or chronic pain conditions restricting exercise
  4. pulmonary or renal failure
  5. active cancer
  6. poorly controlled hypertension (>160/100) or diabetes mellitis (fasting glucose>180 mg/dl, HbA1C >10%)
* Neurological history of

  1. dementia
  2. receptive or global aphasia that confounds testing and training, operationally defined as unable to follow 2 point commands
  3. cognitive deficits (other than dementia and aphasia, as above)

  (e) non-stroke neuromuscular disorder restricting exercise (eg Parkinson's Syndrome) (f) untreated major depression
* exclusion criteria for MRI scanning (metal implants (e.g. pacemaker), claustrophobia, etc.)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
aerobic capacity (peak VO2) | Baseline (timepoint 0) and after training (3 months)
gait velocity | Baseline (timepoint 0) and after training (3 months)

SECONDARY OUTCOMES:
cortical thickness (MRI) | Baseline (timepoint 0) and after training (3 months)
grey matter density (VBM-MRI) | Baseline (timepoint 0) and after training (3 months)
cerebrovascular reserve capacity (ASL-MRI) | Baseline (timepoint 0) and after training (3 months)